CLINICAL TRIAL: NCT04341662
Title: Early Detection of Postpartum Haemorrhage and Treatment Using the World Health Organisation MOTIVE 'First Response' Bundle: a Cluster Randomised Trial With Health Economic Analysis and Mixed-methods Evaluation (E-MOTIVE Trial)
Brief Title: A Clinical Trial to Study the Effectiveness of a Care Bundle to Prevent Bleeding After a Woman Has Given Birth
Acronym: E-MOTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University College, London (Other); University of Melbourne (Other); University of California (Other); World Health Organization (Other); King's College London (Other); University of Liverpool (Other); Jhpiego (Other); Concept Foundation (Other); University of Nairobi (Other); University of Cape Town (Other); Bayero University Kano, Nigeria (Other); Muhimbili University of Health and Allied Sciences (Other); University of Witwatersrand, South Africa (Other); Ammalife (Industry); Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_19-231; PACTR202002791391791 (Registry Identifier: Pan African Clinical Trial Registry)
Record Dates: First submitted 2020-02-07; First posted 2020-04-10 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Post-Partum Haemorrhage
Keywords: post-partum haemorrhage; early detection; blood loss measurement; oxytocin; tranexamic acid
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Parallel cluster randomised trial with a baseline control phase, along with mixed-methods and health economic evaluations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-MOTIVE intervention (Experimental): The E-MOTIVE intervention consists of three elements: 1) a strategy for early detection of PPH, which allows triggering of the 'first response' treatment bundle; 2) a 'first response' bundle called "MOTIVE", based on the WHO guideline recommendations and consisting of uterine Massage, Oxytocic drugs, Tranexamic acid, IV fluids and Examination & Escalation; and 3) an implementation strategy, focusing on simulation-based training with peer-assisted learning, local E-MOTIVE champions, feedback of actionable data to providers, calibrated drape with trigger line, and MOTIVE emergency trolley and/or carry case.
  Interventions: Behavioral: E-MOTIVE intervention
- Usual care (Active Comparator): Usual care with dissemination of the current guidelines
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: E-MOTIVE intervention — The E-MOTIVE intervention consists of three elements: 1) a strategy for early detection of PPH, which allows triggering of the 'first response' treatment bundle; 2) a 'first response' bundle called "MOTIVE", based on the WHO guideline recommendations and consisting of uterine Massage, Oxytocic drugs, Tranexamic acid, IV fluids and Examination & Escalation; and 3) an implementation strategy, focusing on simulation-based training with peer-assisted learning, local E-MOTIVE champions, feedback of actionable data to providers, calibrated drape with trigger line, and MOTIVE emergency trolley and/or carry case.
  Arms: E-MOTIVE intervention
Behavioral: Usual care — Health facilities will continue to follow usual care as per the baseline period for the remainder of the intervention phase.
  Arms: Usual care

SUMMARY:
Every six minutes a mother dies from postpartum haemorrhage (PPH) in low-resource countries, in the prime of her life and often leaving behind a young family. In many settings, when a mother dies in childbirth, her infant has less than a 20% chance of surviving past the first month. PPH, defined as a blood loss of more than 500 ml, is the leading cause of maternal death worldwide, accounting for 27% of maternal deaths. The WHO published "Recommendations for the Prevention and Treatment of Postpartum Hemorrhage" in 2012 to provide evidence-informed recommendations for managing PPH. However, adherence to these recommendations is currently limited by a number of challenges.

This primary aim of this multi-country, parallel cluster randomised trial with a baseline control phase, along with mixed-methods and health economic evaluations, is to evaluate the implementation of early detection and the use of the World Health Organisation (WHO) MOTIVE 'first response' treatment bundle for postpartum haemorrhage (PPH) on clinical, implementation and resource use outcomes. The investigators will evaluate the implementation through mixed-methods and carry out a health economic evaluation from the public healthcare system perspective.

DETAILED DESCRIPTION:
The aim of this trial is evaluate the implementation of early detection and the use of the WHO MOTIVE 'first response' treatment bundle for PPH on clinical, implementation and resource use outcomes. The investigators will evaluate the implementation through mixed-methods and carry out a health economic evaluation from the public healthcare system perspective. The investigators will use a multi-country, parallel cluster randomised trial design with a baseline control phase, along with mixed-methods and health economic evaluations. The trial is conducted in secondary level health facilities in four low- and middle- income countries. For this trial, the health facility is the randomisation unit. Health facilities are eligible for inclusion if they have 1000 to 5000 births a year and provide comprehensive obstetric care with ability to perform surgery for PPH. Pre-existing implementation of early detection or bundled approach are exclusion criteria. The research participants are all healthcare providers attending vaginal births in the study facilities. The E-MOTIVE intervention consists of three elements: 1) a strategy for early detection of PPH, which allows triggering of the 'first response' treatment bundle; 2) a 'first response' bundle called "MOTIVE", based on the WHO guideline recommendations and consisting of uterine Massage, Oxytocic drugs, Tranexamic acid, IV fluids and Examination & Escalation; and 3) an implementation strategy, focusing on simulation-based training with peer-assisted learning, local E-MOTIVE champions, feedback of actionable data to providers, calibrated drape with trigger line, and MOTIVE emergency trolley and/or carry case. The control health facilities will deliver usual care with dissemination of the current guidelines.

The primary outcome is a composite of the following three clinical outcomes: 1) primary severe PPH defined as blood loss ≥1000 ml following a vaginal birth in the facility measured up to 2 hours postpartum; 2) postpartum laparotomy for bleeding until discharge from the health facility; and 3) postpartum maternal death from bleeding until discharge from the health facility. If any of the components occur, this will be deemed as positive for the primary outcome.

The key secondary implementation outcomes of special interest are 1) PPH detection (with the following numerator and denominator: women who objectively had PPH (source-verified blood loss ≥ 500 mL after weighing of the drape) and were diagnosed with PPH by the birth attendants divided by the total number of women who objectively had PPH (source verified blood loss ≥ 500 mL after weighing the drape), and 2) compliance with MOTIVE bundle (with the following numerator and denominator: women who objectively had PPH and were treated with the PPH bundle following a diagnosis of PPH by the birth attendants divided by the total number of women who objectively had PPH (blood loss ≥ 500 mL after weighing of the drape).

Secondary outcomes: blood transfusion, uterine tamponade, Intensive Care Unit admissions or higher-level facility transfers, and new-born deaths along with implementation and resource use outcomes.

Eighty health facilities will take part in the study. Initially, all health facilities will enter a 7-month baseline period in which they will be following usual care. After this, we will randomise 40 of the 80 health facilities to the E-MOTIVE intervention for 7 months, allowing two months for transition. The other 40 health facilities will continue to follow usual care as per the baseline period for the entire trial duration (16 months). The anticipated sample size for the study will be 215,040 women. This sample size is expected to have over 90% power to detect a 25% relative reduction in the primary outcome from 4% to 3% after allowing for clustering. The number of clusters has been inflated by 10% to allow for drop out of health facilities and for varying cluster sizes. Randomisation will use a minimisation algorithm to balance the intervention and control facilities by the number of vaginal births per health facility, the health facility rate of the composite primary outcome during the baseline phase, the quality of oxytocin used per health facility, and the number of facilities in each arm.

During the 7-month baseline phase, the investigators will refine and optimise the E-MOTIVE implementation strategy by piloting it in two to three facilities per country over up to two adaptive cycles for addressing barriers and enablers to delivery and implementation, ahead of the intervention phase.

The investigators will also conduct a mixed-methods process evaluation to assess the extent to which the E-MOTIVE intervention has been implemented as intended. The implementation outcomes of interest are fidelity, adoption, adaptation, acceptability, and sustainability, as well as contextual influences and barriers and enablers to implementation.

The investigators plan to assess the cost-effectiveness of the E-MOTIVE intervention compared with usual care from a public healthcare system perspective for each country, as measured by incremental cost-effectiveness ratios for a) severe PPH prevented, b) laparotomy for PPH prevented, c) death from PPH avoided, and (d) quality-adjusted life-years prevented.

Following the publication of the E-MOTIVE trial findings, a prospective pre-post intervention study of the E-MOTIVE intervention was planned in eight secondary-level care District Head Quarter (DHQ) hospitals in the Sindh and Punjab provinces of Pakistan. Pakistan was originally scheduled to be part of the multi-country, cluster-randomised E-MOTIVE trial. However, the catastrophic floods in Pakistan in 2022 delayed the start of recruitment, whilst the other participating countries progressed to complete the trial. At this stage, as the required sample size for the trial had been achieved, the Independent Data Monitoring Committee advised completing and analysing the trial without the participation of Pakistan. The definitive effects found by the E-MOTIVE trial made it unethical to conduct further randomised trials of the intervention. As all countries that contributed to the E-MOTIVE trial were from Africa, an outstanding question on generalisability of the findings outside of Africa remained. The E-MOTIVE study in Pakistan was, therefore, planned as a pre-post study to assess the implementation and generalisability of E-MOTIVE in a South Asian healthcare setting. The amended protocol was approved by the University of Birmingham, UK and the Pakistan ethics and regulatory review committee. The study retained the same primary clinical and implementation outcomes as the main trial.

ELIGIBILITY:
Cluster: Health facility is the randomisation unit. Health facilities are eligible for inclusion if they have 1000 to 5000 births a year and provide comprehensive obstetric care with ability to perform surgery for PPH. Health facilities are selected based on being administratively and geographically distinct from each other. Pre-existing implementation of early detection or bundled approach are exclusion criteria

Research participants: All healthcare providers attending vaginal births at the study facilities.

Patients: All verified vaginal births in the study facilities

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99659 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arri Coomarasamy, MD, Principal Investigator — University of Birmingham
Locations (6):
- University of Nairobi, Nairobi, Kenya
- Bayero University, Kano, Nigeria
- Aga Khan University, Karachi, Pakistan
- South Africa (2):
  - University of Cape Town, Cape Town
  - University of the Witwatersrand, Johannesburg
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after primary publication
Access Criteria: Data sharing will be subject to agreement by the Trial Management Group
URL: http://www.birmingham.ac.uk/emotive

REFERENCES:
- [Result] Gallos I, Devall A, Martin J, Middleton L, Beeson L, Galadanci H, Alwy Al-Beity F, Qureshi Z, Hofmeyr GJ, Moran N, Fawcus S, Sheikh L, Gwako G, Osoti A, Aswat A, Mammoliti KM, Sindhu KN, Podesek M, Horne I, Timms R, Yunas I, Okore J, Singata-Madliki M, Arends E, Wakili AA, Mwampashi A, Nausheen S, Muhammad S, Latthe P, Evans C, Akter S, Forbes G, Lissauer D, Meher S, Weeks A, Shennan A, Ammerdorffer A, Williams E, Roberts T, Widmer M, Oladapo OT, Lorencatto F, Bohren MA, Miller S, Althabe F, Gulmezoglu M, Smith JM, Hemming K, Coomarasamy A. Randomized Trial of Early Detection and Treatment of Postpartum Hemorrhage. N Engl J Med. 2023 Jul 6;389(1):11-21. doi: 10.1056/NEJMoa2303966. Epub 2023 May 9. PMID 37158447
- [Derived] Williams EV, Goranitis I, Oppong R, Perry SJ, Devall AJ, Martin JT, Mammoliti KM, Beeson LE, Sindhu KN, Galadanci H, Alwy Al-Beity F, Qureshi Z, Hofmeyr GJ, Moran N, Fawcus S, Mandondo S, Middleton L, Hemming K, Oladapo OT, Gallos ID, Coomarasamy A, Roberts TE. A cost-effectiveness analysis of early detection and bundled treatment of postpartum hemorrhage alongside the E-MOTIVE trial. Nat Med. 2024 Aug;30(8):2343-2348. doi: 10.1038/s41591-024-03069-5. Epub 2024 Jun 6. PMID 38844798
- [Derived] Forbes G, Akter S, Miller S, Galadanci H, Qureshi Z, Fawcus S, Hofmeyr GJ, Moran N, Singata-Madliki M, Dankishiya F, Gwako G, Osoti A, Thomas E, Gallos I, Mammoliti KM, Devall A, Coomarasamy A, Althabe F, Atkins L, Bohren MA, Lorencatto F. Factors influencing postpartum haemorrhage detection and management and the implementation of a new postpartum haemorrhage care bundle (E-MOTIVE) in Kenya, Nigeria, and South Africa. Implement Sci. 2023 Jan 11;18(1):1. doi: 10.1186/s13012-022-01253-0. PMID 36631821
- [Derived] Akter S, Forbes G, Miller S, Galadanci H, Qureshi Z, Fawcus S, Justus Hofmeyr G, Moran N, Singata-Madliki M, Amole TG, Gwako G, Osoti A, Thomas E, Gallos I, Mammoliti KM, Coomarasamy A, Althabe F, Lorencatto F, Bohren MA. Detection and management of postpartum haemorrhage: Qualitative evidence on healthcare providers' knowledge and practices in Kenya, Nigeria, and South Africa. Front Glob Womens Health. 2022 Nov 18;3:1020163. doi: 10.3389/fgwh.2022.1020163. eCollection 2022. PMID 36467287
- [Derived] Bohren MA, Lorencatto F, Coomarasamy A, Althabe F, Devall AJ, Evans C, Oladapo OT, Lissauer D, Akter S, Forbes G, Thomas E, Galadanci H, Qureshi Z, Fawcus S, Hofmeyr GJ, Al-Beity FA, Kasturiratne A, Kumarendran B, Mammoliti KM, Vogel JP, Gallos I, Miller S. Formative research to design an implementation strategy for a postpartum hemorrhage initial response treatment bundle (E-MOTIVE): study protocol. Reprod Health. 2021 Jul 14;18(1):149. doi: 10.1186/s12978-021-01162-3. PMID 34261508
- See also: Trial website — http://www.birmingham.ac.uk/emotive

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Women were excluded from the final analysis if their blood loss data could not be source-verified with photographic evidence of the blood collection drape on the weighing scales (displaying the drape weight) which could be linked to the patient I.D number
Period: Overall Study
Arm/Group | E-MOTIVE Intervention | Usual Care
Started | 49101 (Number of women with a CRF) | 50558 (Number of women with a CRF)
Completed | 48678 (Number of women with record of primary outcome) | 50044 (Number of women with record of primary outcome)
Not Completed | 423 | 514
Not completed — Did not have source-verified blood loss data | 423 | 514

BASELINE CHARACTERISTICS:
Population: The numbers provided are for patients however the participant flow refers to clusters (hospitals)
Groups:
- Total: Total of all reporting groups
Arm/Group | E-MOTIVE Intervention | Usual Care | Total
Number analyzed (Participants) | 49101 | 50558 | 99659
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [21 to 31] | 26 [21 to 30] | 26 [21 to 31]
Sex: Female, Male [Count of Participants; unit: Participants] — Only female patients participated
  Participants
    Female | 49101 | 50558 | 99659
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Tanzania | 10658 | 10627 | 21285
  South Africa | 9668 | 9030 | 18698
  Kenya | 11475 | 9992 | 21467
  Nigeria | 17300 | 20909 | 38209

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is a Composite of the Following Three Clinical Outcomes: 1) Severe PPH Defined as Blood Loss ≥1000 ml or; 2) Postpartum Laparotomy for Bleeding or; 3) Postpartum Maternal Death From Bleeding. Please See Below for Further Details.
Description: 1. Number of women with primary severe PPH defined as blood loss ≥1000 ml following a vaginal birth in the facility up to 2 hours postpartum
  2. Number of women with postpartum laparotomy for bleeding until discharge from the health facility
  3. Number of postpartum maternal deaths from bleeding until discharge from the health facility.
  A Blinded Endpoint Review Committee (BERC) will assess incoming data relevant to the primary outcome in order to confirm if any postpartum laparotomy was performed for bleeding and if any maternal death was due to bleeding
Time Frame: Postpartum until discharge from the health facility (up to 42 days)
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 794 | 2139

2. Secondary Outcome: PPH Detection
Description: With the following numerator and denominator: women who objectively had PPH (source-verified blood loss ≥ 500 mL after weighing of the drape) and were diagnosed with PPH by the birth attendants divided by the total number of women who objectively had PPH (source verified blood loss ≥ 500 mL after weighing the drape)
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 4158 | 8351
Participants | 3,870 | 4,244

3. Secondary Outcome: Compliance With MOTIVE Bundle
Description: Defined as adherence with three core elements of the bundle: administration of oxytocic drugs, TXA and IV fluids. If all three core elements are administered when a PPH is diagnosed, this will be deemed positive for bundle compliance
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 4158 | 8351
Participants | 3791 | 1623

4. Secondary Outcome: Number of Women With Laparotomy Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days)
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 13 | 9

5. Secondary Outcome: Number of Women With Laparotomy With Compression Sutures Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 1 | 1

6. Secondary Outcome: Number of Women With Laparotomy With Arterial Ligation Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the healthcare facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 0 | 2

7. Secondary Outcome: Number of Women With Hysterectomy Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 11 | 6

8. Secondary Outcome: Number of Women With Hysterectomy for Bleeding Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 9 | 6

9. Secondary Outcome: Rate of All Cause Maternal Mortality Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 17 | 28

10. Secondary Outcome: Amount of Blood Loss (as a Continuous Variable)
Description: Reported in millilitres
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Median (Inter-Quartile Range); unit: Millilitres
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Millilitres | 160 [100 to 280] | 220 [120 to 380]

11. Secondary Outcome: Number of Women With Primary PPH Defined as Blood Loss ≥500 ml
Description: Measured in mililitres
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 4,158 | 8,351

12. Secondary Outcome: Duration of Hospitalisation Postpartum
Description: Measured in days
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Days | 1 [0 to 1] | 1 [0 to 1]

13. Secondary Outcome: Duration of ICU Hospitalisation Postpartum
Description: Measured in days
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Days | 1 [0 to 3] | 1 [1 to 2]

14. Secondary Outcome: Number of Women Transferred to a Higher-level Facility Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 85 | 18

15. Secondary Outcome: Rate of All Cause Neonatal Mortality Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49923 | 51535
Participants | 2259 | 2233

16. Secondary Outcome: Number of Women Receiving Non-pneumatic Anti-shock Garment (NASG) Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 90 | 38

17. Secondary Outcome: Number of Women Receiving Uterine Balloon Tamponade Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 44 | 57

18. Secondary Outcome: Number of Women Receiving a Blood Transfusion Postpartum Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 1074 | 1296

19. Secondary Outcome: Number of Women Receiving Blood Transfusion for Postpartum Haemorrhage Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 580 | 944

20. Secondary Outcome: Number of Women Admitted to Intensive Care Unit (ICU) Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 7 | 32

21. Secondary Outcome: Number of Women With Primary Severe PPH (Defined as Blood Loss ≥1000 ml) Following a Vaginal Birth in the Facility Measured up to 2 Hours Postpartum
Time Frame: Up to 2 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 786 | 2,129

22. Secondary Outcome: Postpartum Laparotomy for Bleeding Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 12 | 7

23. Secondary Outcome: Postpartum Maternal Death From Bleeding Until Discharge From the Health Facility
Time Frame: Postpartum until discharge from the health facility (up to 42 days).
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 12 | 18

24. Secondary Outcome: PPH Treatment by Healthcare Provider up to 2 Hours Postpartum (or up to 24 Hours if Bleeding Continues)
Description: With the following numerator and denominator: women diagnosed with PPH by the birth attendants divided by the total of women having a vaginal birth in the health facility
Time Frame: Up to 2 hours postpartum (or up to 24 hours if bleeding continues)
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 5921 | 4899

25. Secondary Outcome: Bundle Usage up to 2 Hours Postpartum (or up to 24 Hours if Bleeding Continues)
Description: With the following numerator and denominator: women treated with the PPH bundle following a diagnosis of PPH by the birth attendants divided by the total of women having a vaginal birth in the health facility
Time Frame: Up to 2 hours postpartum (or up to 24 hours if bleeding continues)
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 49101 | 50558
Participants | 5,783 | 1,725

26. Secondary Outcome: Bundle Usage for PPH up to 2 Hours Postpartum (or up to 24 Hours if Bleeding Continues)
Description: With the following numerator and denominator: women treated with the PPH bundle following a diagnosis of PPH by the birth attendant divided by the total of women diagnosed with PPH by the birth attendants
Time Frame: Up to 2 hours postpartum (or up to 24 hours if bleeding continues)
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 5783 | 1725

27. Secondary Outcome: Number of Women Receiving Uterine Massage for PPH
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 5794 | 4119

28. Secondary Outcome: Number of Women Receiving Oxytocin for PPH
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 5897 | 4321

29. Secondary Outcome: Number of Women Receiving Misoprostol for PPH
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 2601 | 2732

30. Secondary Outcome: Number of Women Receiving TXA for PPH
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 5829 | 1983

31. Secondary Outcome: Number of Women Receiving Intravenous Fluids (IV) for PPH
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 5884 | 4199

32. Secondary Outcome: Number of Women Receiving Examination of the Genital Tract
Description: Physical observation (no specific tool used).
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 5506 | 3608

33. Secondary Outcome: Number of Women Receiving Any Treatment Uterotonic for PPH
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 5909 | 4541

34. Secondary Outcome: Number of Women Requiring Additional Treatment Interventions (Not Responding to the MOTIVE Bundle).
Time Frame: Up to 24 hours postpartum
Population: Number of women
Measure: Count of Participants; unit: Participants
Arm/Group | E-MOTIVE Intervention | Usual Care
Number analyzed (Participants) | 5921 | 4899
Participants | 219 | 637

ADVERSE EVENTS:
Time Frame: As the interventions being tested as a bundle in this trial are recommended and used throughout the world, there are no adverse events which would be anticipated as a unique consequence of participation in the trial. No expedited reporting of adverse events is proposed. Maternal deaths and ICU admissions were collected until discharge from the health facility (up to 42 days)
Arm/Group | E-MOTIVE Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 17/49101 | 28/50558
Serious Adverse Events (participants affected / at risk) | 7/49101 | 32/50558
Other Adverse Events (participants affected / at risk) | 0/49101 | 0/50558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-MOTIVE Intervention (N=49101) | Usual Care (N=50558)
Admission to ICU (Pregnancy, puerperium and perinatal conditions) | 7 | 32 — Intensive Care Unit (ICU) admission postpartum until discharge from the health facility

LIMITATIONS AND CAVEATS:
Study limitations include the lack of certain secondary outcomes such as post-natal hemoglobin level and anemia rates, and women's experience of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT04341662/Prot_002.pdf
  • Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04341662/SAP_001.pdf